CLINICAL TRIAL: NCT06854536
Title: A Study on the Changes and Prognosis of Intestinal Microbiota and Function in Infants With Food Allergies
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GMSF-001
Record Dates: First submitted 2025-02-08; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Health; Children; Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Food-allergic children: Children diagnosed with food allergies

SUMMARY:
Microorganisms maintain a complex interrelationship with the human body, influencing each other. In recent years, people have gradually realized that the formation of the pediatric microecosystem is closely related to the development of gastrointestinal and even systemic immunity in children. The establishment of the pediatric microecosystem during childhood has significant implications for various diseases in adulthood. They are crucial for the host's nutrition, metabolism, resistance to pathogens, and immune function. Increasing evidence supports the association between gut microbiota abnormalities and the pathophysiology of food allergies, but the conclusions of existing clinical efficacy studies remain controversial. Previous research by the team has found that the gut microbiome has a clear impact on the occurrence and development of digestive and allergic diseases in children.

DETAILED DESCRIPTION:
Food allergy is a harmful immunological response to the ingestion of food proteins , causing various symptoms in multiple parts of the body, such as skin itching, redness, and hives; asthma and coughing in the respiratory tract; and nausea, vomiting, and diarrhea in the gastrointestinal tract. In severe cases, it can even lead to shock and death. FA primarily affects infants and young children, with a prevalence rate of up to 10% in developed countries. A epidemiological survey in China showed that the food allergy rate among children aged 0-36 months in eight cities was 6.53%, and the incidence rate has been increasing year by year. Currently, it is believed that FA in infancy is a risk factor for later eczema, allergic rhinitis, and asthma, which can severely impact children's growth and development and quality of life, increasing the burden on families and society. It has become a public health issue worldwide. Among infant food allergies, cow's milk and egg allergies are the most common. Cow's milk protein is the most commonly used protein source in ordinary infant formulas. Cow's milk protein allergy refers to an adverse reaction mediated by the immune mechanism caused by the body's response to cow's milk protein, which can be mediated by IgE, non-IgE, or both. Studies in some Chinese cities have shown that the prevalence of Cow's milk protein allergy among infants aged 0-3 years is approximately 0.83% to 3.5%. Since cow's milk protein is essential for infant growth and development, Cow's milk protein allergy can significantly affect children's growth and development and quality of life.

The pathogenesis of FA is not yet fully understood, but increasing evidence supports the involvement of abnormal gut microbiota in the pathophysiology of FA. Extensive basic research has found that certain probiotics play roles at multiple stages in the development of food allergies, including: In the intestinal lumen: regulating the structure of gut microbiota, increasing the production of secretory IgA, and modifying antigen peptides. At the intestinal mucosal level: improving intestinal mucosal permeability, stimulating the growth and differentiation of intestinal epithelial cells. At the submucosal level: regulating the function of the innate and adaptive immune systems, inducing oral tolerance, and affecting the function of the enteric neuroendocrine system. Studies have shown that bifidobacteria in the host gut can promote the development and maturation of the infant immune system, and their species composition and diversity have received significant attention regarding their impact on allergic diseases.

In summary, food allergies are relatively common in infancy and have been increasing annually. Therefore, this study aims to understand the changes in the gut microbiota and its metabolites in infants with food allergies, as well as the differences in gut microbiota between children with and without immune tolerance to food allergies, and to discover related gut microbial metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-36 months old
* Both men and women;
* The child's legal guardian signed the informed consent to participate in the study.
* The legal guardian of the child commits to follow the study procedures and cooperate with the entire study process

Exclusion Criteria:

* Probiotics or antibiotics within 1 month
* Associated with clinically significant abnormalities in liver and kidney function, nervous system, respiratory system, and coagulation function as determined by the investigator
* Unstable vital signs;
* Have other underlying medical conditions
* Individuals deemed unsuitable for this clinical trial.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Diagnosed with food allergy children aged 1-36 months old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiome analysis | The time point of confirming food allergy and the age of 36 months
  The fecal samples from all participants will be collected and subjected to high-throughput metagenomic sequencing in order to elucidate the characteristics and composition of the intestinal microbiome in children with food allergies.
Intestinal microbiome metabolites analysis | The time point of confirming food allergy and the age of 36 months
  This will be detected and analyzed by liquid chromatography-mass spectrometry (LC-MS) non-targeted metabolomics to analyze the metabolites of the intestinal microbiome.

SECONDARY OUTCOMES:
Differences in clinical symptoms | 36 months of age
  The incidence of ariway allergy in children with food allergy at the age of 36 months.
The percentile number of height of children at different groups | The time point of confirming food allergy and the age of 36 months
  Compare the Percentile number of height of children with diagnosed with food allergy and healthy children.
The percentile number of head circumference of children at different group | The time point of confirming food allergy and the age of 36 months
  Compare the Percentile number of head circumference of children with diagnosed with food allergy and healthy children.
The percentile number of weight of children at different groups | The time point of confirming food allergy and the age of 36 months
  Compare the Percentile number of weight of children with diagnosed with food allergy and healthy children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China